CLINICAL TRIAL: NCT05865834
Title: Effectiveness of E-health Intervention Using Smart Phone App to Reduce Anxiety & Depressive Symptoms Among Adolescents: A Cluster Randomized Controlled Trial
Brief Title: Improvement of Mental Health in Adolescents Using E-health Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Shafquat Rozi, Assistant Professor/ Director of MSc. Epidemiology and Biostatistics, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 8053
Record Dates: First submitted 2023-05-08; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Mental Disorder in Adolescence; Depression in Adolescence; Anxiety Disorders
Keywords: Mental health; anxiety; depression; e-heath intervention; mental health application; adolescents
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being; Depression

STUDY DESIGN:
Intervention Model Description: A two-stage cluster sampling will be employed. Randomization will occur at school level for 2 arms i.e. interventional and control groups. Students will be selected randomly from each group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm (Experimental): One public and one private school will be randomly placed into intervention arm. Students from grade 6th - grade 10th will be recruited on their willingness to participant.
  A smartphone application will be installed on the personal gadgets of the students in the interventional arm at baseline. For assessing the effectiveness of this app, the first follow-up will be done at one month after the intervention and the second follow up after 3 months to evaluate whether the application had an impact on their depressive and anxiety symptom using PHQ-A, GAD-7 and WHO-5 scales.
  Interventions: Other: A smartphone application
- control arm (Active Comparator): one public and one private school will be randomly allocated to control arm. Students from grade 6th - grade 10th will be recruited on their willingness to participant.
  the control group will receive self-reading educational leaflets. the first follow-up will be done at one month after the intervention and the second follow up after 3 months to evaluated whether the application had an impact on their depressive and anxiety symptom using PHQ-A, GAD-7 and WHO-5 scales.
  Interventions: Other: Pictorial educational leaflets

INTERVENTIONS:
Other: A smartphone application — app will have 2 modules: Chill zone and sleep; Chill zone has 9 sub-modules which are meditation, breathing techniques, family time, art time, funny sayings, reframe stress and relax, diet and cooking tips, mini courses and how to become better. The sub-modules of sleep are: wind down, sleep music, storytelling, nature sounds and beautiful nature. These modules will be approved by a clinical psychologist to help people with symptoms of depression and anxiety. Skills learned include emotion recognition, emotional management, behavioral activation (being active), recognizing and challenging unhelpful thoughts and cognitive restructuring to plan for their future.
  Arms: intervention arm
Other: Pictorial educational leaflets — the control group will receive self-reading educational leaflets, the majority of which are pictorial. These leaflets will be approved by a clinical psychologist to help people with symptoms of depression and anxiety.
  Arms: control arm

SUMMARY:
the goal of this cluster randomized controlled trial is to assess the effectiveness of smartphone application in reducing the symptoms of Anxiety and depression among adolescents. The main objectives of this trial are:

1. Primary Objective To develop a smart phone application for reduction in depressive and anxiety symptoms in Pakistani adolescents aged 12-18 years
2. Secondary Objectives

   * To determine the effectiveness of a smart phone application in reduction of anxiety symptoms in Pakistani adolescents aged 12-18 years via a randomized controlled trial
   * To determine the effectiveness of a smart phone application in reduction of depressive symptoms in Pakistani adolescents aged 12-18 years via a randomized controlled trial
   * To determine the effectiveness of a smart phone application in improvements of well-being of Pakistani adolescents aged 12-18 years via a randomized controlled trial

the randomization will occur at the school level for the intervention group and control group.

Students in the intervention group will receive the access to a smartphone application designed to improve the mental health of adolescents, they will be briefed on how to use the application and its advantages. while the students in the control group will receive self-reading pictorial educational leaflets related to mental health improvement.

the researcher will conduct the assessment of depression, anxiety and mental wellbeing using PHQ-A, GAD-7 and WHO-5 at baseline, 1 month and at 3 months to compare if the smartphone application is effective in reducing the symptoms of depression and anxiety of adolescents and overall improvement in the mental wellbeing.

DETAILED DESCRIPTION:
As per World Health Organization (WHO), 13% of adolescents worldwide experience a mental disorder. Also, depression, anxiety, and other behavioral disorders are leading causes of mortality and disability in this age bracket. The advent of the pandemic has further worsened the mental health situation in adolescents. If the increasing burden of mental health issues is not addressed in adolescence, they can culminate into established mental disorders extending to adulthood, impairing overall wellbeing and limiting opportunities. In order to cater to mental health issues in adolescents at an early stage, we aim to develop a smartphone application for the reduction of depression and anxiety symptoms in school-going adolescents aged 12-18 years.

Also, we plan to assess the effectiveness of the smartphone application via a cluster randomized controlled trial. The curated smartphone application will have two modules: Chill zone and sleep; Chill zone will comprise of 9 sub-modules and sleep 5 sub-modules. The 9 sub-modules of the Chill zone will be as follows; meditation, breathing techniques, family time, art time, funny sayings, reframe stress and relax, diet and cooking tips, mini-courses, and how to become better. The sub-modules of sleep will be winding down, sleep music, storytelling, nature sounds, and beautiful nature. Each module will be designed to be completed on separate days with daily push notifications.

Once the application is designed, the trial will be conducted in schools of Karachi. The intervention and control arm will have two schools with 50 students/school from grades 6-10. The total sample size will be 200 students. A two-stage cluster sampling with stratification on school type (government or private) will be employed to select schools and recruit students. Participants allocated to the intervention arm will be given mental health intervention, and the students in the control arm will be given educational leaflets. PHQ-A, GAD-7, and WHO depression wellbeing scale for assessing depressive symptoms, anxiety symptoms, and wellbeing will be used at baseline, 1 month, and three months. Generalized estimating equation, will be used to compare mean scores of depression, anxiety and wellbeing scores between both arms.

ELIGIBILITY:
Inclusion Criteria:

* Registered secondary schools with the Board of Secondary Education Karachi who will provide consent to participate in the study
* 12-18-year-olds adolescents enrolled in public and private school of Karachi Pakistani
* The intervention and control arm must understand English or Urdu in order to use the mobile-based application.
* Intervention group must have access to a smartphone or portable smart device (Electronic Tablets, iPad, etc.).
* Participants having access to Wi-Fi at home- or on the phone for downloading the app.
* Parenteral consent is required for an adolescent to participate in this study; simultaneously, an individual's consent is equally important to be included in this trial.
* Moreover, students will be asked to participate in the study if they:(a) experience mild to moderate depression defined as scoring above the cut-off score of 4 on the Patient Health Questionnaire for adolescents (PHQ-A) and/or anxiety symptoms defined as scoring above the cut-off score of 5 on the Generalized Anxiety Disorder scale-7 items (GAD-7 (b) had a well-being score of ≤50 on World Health Organization Well-Being scale (WHO-5) at basic screening level.

Exclusion Criteria:

* School authorities who did not grant permission to conduct the research study in their school
* School unable or unwilling to provide informed consent /assent
* students not willing to participate in the study
* Use of a mobile device that does not comply with the app requirements (non- android phone holders)
* Have no internet access or smartphone
* Students will be excluded if they: (a) any chronic disease (c) currently taking psychiatric consultation/ treatment for depression/ anxiety, or have received treatment/therapy in the past 12 months

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Anxiety | 6 months
  change in the level of anxiety symptoms using the Generalized anxiety scale (GAD-7)
Depression | 6 months
  Change in the level of depressive symptoms assessed using Patient Health Questionnaire (PHQ-A) adapted for adolescents
Mental well-being | 6 months
  change in the mental well-being scores assessed using WHO-5 scale

CONTACTS AND LOCATIONS:
Overall Officials: Shafquat Rozi, Ph D., Principal Investigator — Aga Khan Hospital -Karachi
Locations (1):
- Aga Khan University- Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balaji M, Andrews T, Andrew G, Patel V. The acceptability, feasibility, and effectiveness of a population-based intervention to promote youth health: an exploratory study in Goa, India. J Adolesc Health. 2011 May;48(5):453-60. doi: 10.1016/j.jadohealth.2010.07.029. Epub 2010 Oct 2. PMID 21501803
- [Background] Dawson KS, Watts S, Carswell K, Shehadeh MH, Jordans MJD, Bryant RA, Miller KE, Malik A, Brown FL, Servili C, van Ommeren M. Improving access to evidence-based interventions for young adolescents: Early Adolescent Skills for Emotions (EASE). World Psychiatry. 2019 Feb;18(1):105-107. doi: 10.1002/wps.20594. No abstract available. PMID 30600639
- [Background] Day V, McGrath PJ, Wojtowicz M. Internet-based guided self-help for university students with anxiety, depression and stress: a randomized controlled clinical trial. Behav Res Ther. 2013 Jul;51(7):344-51. doi: 10.1016/j.brat.2013.03.003. Epub 2013 Mar 28. PMID 23639300
- [Background] de Bruin EJ, Bogels SM, Oort FJ, Meijer AM. Efficacy of Cognitive Behavioral Therapy for Insomnia in Adolescents: A Randomized Controlled Trial with Internet Therapy, Group Therapy and A Waiting List Condition. Sleep. 2015 Dec 1;38(12):1913-26. doi: 10.5665/sleep.5240. PMID 26158889
- [Background] Gao Y, Li LP, Kim JH, Congdon N, Lau J, Griffiths S. The impact of parental migration on health status and health behaviours among left behind adolescent school children in China. BMC Public Health. 2010 Feb 3;10:56. doi: 10.1186/1471-2458-10-56. PMID 20128901
- [Background] Ha T, van Roekel E, Iida M, Kornienko O, Engels RCME, Kuntsche E. Depressive Symptoms Amplify Emotional Reactivity to Daily Perceptions of Peer Rejection in Adolescence. J Youth Adolesc. 2019 Nov;48(11):2152-2164. doi: 10.1007/s10964-019-01146-4. Epub 2019 Oct 16. PMID 31620972
- [Background] Hellfeldt K, Lopez-Romero L, Andershed H. Cyberbullying and Psychological Well-being in Young Adolescence: The Potential Protective Mediation Effects of Social Support from Family, Friends, and Teachers. Int J Environ Res Public Health. 2019 Dec 19;17(1):45. doi: 10.3390/ijerph17010045. PMID 31861641
- [Background] Karyotaki E, Klein AM, Riper H, Wit L, Krijnen L, Bol E, Bolinski F, Burger S, Ebert DD, Auerbach RP, Kessler RC, Bruffaerts R, Batelaan N, van der Heijde CM, Vonk P, Kleiboer A, Wiers RW, Cuijpers P. Examining the effectiveness of a web-based intervention for symptoms of depression and anxiety in college students: study protocol of a randomised controlled trial. BMJ Open. 2019 May 14;9(5):e028739. doi: 10.1136/bmjopen-2018-028739. PMID 31092668
- [Background] Khalid A, Qadir F, Chan SWY, Schwannauer M. Adolescents' mental health and well-being in developing countries: a cross-sectional survey from Pakistan. J Ment Health. 2019 Aug;28(4):389-396. doi: 10.1080/09638237.2018.1521919. Epub 2018 Nov 19. PMID 30451053
- [Background] Mason-Jones AJ, Crisp C, Momberg M, Koech J, De Koker P, Mathews C. A systematic review of the role of school-based healthcare in adolescent sexual, reproductive, and mental health. Syst Rev. 2012 Oct 26;1:49. doi: 10.1186/2046-4053-1-49. PMID 23098138
- [Background] Moore SE, Norman RE, Suetani S, Thomas HJ, Sly PD, Scott JG. Consequences of bullying victimization in childhood and adolescence: A systematic review and meta-analysis. World J Psychiatry. 2017 Mar 22;7(1):60-76. doi: 10.5498/wjp.v7.i1.60. eCollection 2017 Mar 22. PMID 28401049
- [Background] Rao S, Shah N, Jawed N, Inam S, Shafique K. Nutritional and lifestyle risk behaviors and their association with mental health and violence among Pakistani adolescents: results from the National Survey of 4583 individuals. BMC Public Health. 2015 Apr 28;15:431. doi: 10.1186/s12889-015-1762-x. PMID 25927931
- [Background] Razzak HA, Harbi A, Ahli S. Depression: Prevalence and Associated Risk Factors in the United Arab Emirates. Oman Med J. 2019 Jul;34(4):274-282. doi: 10.5001/omj.2019.56. PMID 31360314
- [Background] Salam RA, Das JK, Lassi ZS, Bhutta ZA. Adolescent Health and Well-Being: Background and Methodology for Review of Potential Interventions. J Adolesc Health. 2016 Oct;59(4S):S4-S10. doi: 10.1016/j.jadohealth.2016.07.023. PMID 27664594
- [Background] van Dalen M, Dierckx B, Pasmans SGMA, Aendekerk EWC, Mathijssen IMJ, Koudstaal MJ, Timman R, Williamson H, Hillegers MHJ, Utens EMWJ, Okkerse JME. Anxiety and depression in adolescents with a visible difference: A systematic review and meta-analysis. Body Image. 2020 Jun;33:38-46. doi: 10.1016/j.bodyim.2020.02.006. Epub 2020 Feb 21. PMID 32092507
- [Background] Zisk A, Abbott CH, Bounoua N, Diamond GS, Kobak R. Parent-teen communication predicts treatment benefit for depressed and suicidal adolescents. J Consult Clin Psychol. 2019 Dec;87(12):1137-1148. doi: 10.1037/ccp0000457. Epub 2019 Oct 24. PMID 31647277
- [Background] Grist R, Porter J, Stallard P. Mental Health Mobile Apps for Preadolescents and Adolescents: A Systematic Review. J Med Internet Res. 2017 May 25;19(5):e176. doi: 10.2196/jmir.7332. PMID 28546138